CLINICAL TRIAL: NCT03614429
Title: Management of Urethral Injury During Penile Prosthesis Implantation: Urethral Sterilization With Chlorhexidine Digluconate to Facilitate Primary Repair and Same-Session Implantation
Brief Title: Urethral Sterilization With Chlorhexidine Digluconate to Facilitate Primary Repair & Same-Session Implantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Osama Kamal Shaeer, Professor of Andrology, Sexual Medicine & STDs, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1-4-2018
Record Dates: First submitted 2018-07-29; First posted 2018-08-03 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Penile Prosthesis; Complications
Keywords: Penile Prosthesis; Urethral injury; Urethral sterilization

STUDY DESIGN:
Intervention Model Description: Comparative experimental (interventional) controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Group 1: control group, n=50 Male patients undergoing aseptic surgery (regardless the procedure)
  Inclusion criteria Male patients aged 20-50 years-old or older undergoing a sterile surgical procedure.
  Exclusion criteria Unwilling patient for this procedure Patients with history of urethral surgery, urinary calculi, urethral structure, or ongoing pyospermia, prostatitis or pyuria will be excluded, and so will be patients undergoing non-sterile surgeries such as abscess drainage.
- Ch group (Experimental): Group 2: Chlorhexidine group (Ch group), n=50 Male patients undergoing aseptic surgery (regardless the procedure)
  Inclusion criteria Male patients aged 20-50 years-old or older undergoing a sterile surgical procedure.
  Exclusion criteria Unwilling patient for this procedure Patients with history of urethral surgery, urinary calculi, urethral structure, or ongoing pyospermia, prostatitis or pyuria will be excluded, and so will be patients undergoing non-sterile surgeries such as abscess drainage.
  Interventions: Drug: Chlorhexidine gel will be prepared according to an international product Instillagel®

INTERVENTIONS:
Drug: Chlorhexidine gel will be prepared according to an international product Instillagel® — Pre-operatively, urethral instillation with Chlorhexidine gel will be performed for the Ch group, while for the control group, instillation will not be performed.
  Chlorhexidine gel will be prepared according to an international product; Instillagel®, used prior to urethral catheterization as analgesic / anti-septic, with the following composition:
  6ml of Instillagel® gel contain: 117.6mg lidocaine hydrochloride, 3.1mg chlorhexidine digluconate, 3.8mg methyl hydroxybenzoate (E218), 1.6mg propyl hydroxybenzoate (E216) 11ml of Instillagel® gel contain: 215.7mg lidocaine hydrochloride, 5.8mg chlorhexidine digluconate, 6.9mg methyl hydroxybenzoate (E218), 2.9mg propyl hydroxybenzoate (E216)
  The other ingredients are:
  Hyetellose, propylene glycol* (E 1520), sodium hydroxide and purified water. Intra-operatively, the Ch group will receive Chlorhexidine instillation again before surgery, while the control group will not.
  Arms: Ch group

SUMMARY:
The introduction of penile implants has revolutionized the management of male erectile dysfunction. However, a number of intraoperative complications may occur, which have a major impact on clinical outcomes and patient satisfaction such as bleeding, infection and urethral injury.

Patients undergoing penile implant surgery with fibrotic corpora (e.g., after priapism, after infection, or with Peyronie disease) have a higher risk rates of urethral perforation. This may be related to previous scarring, the difficultly in dilating scarred and fibrotic corpora and its inherent risk of corporal crossover and urethral perforation.

This work examines the efficacy of pre-operative urethral sterilization in rendering the urethra as sterile as the skin of the genital area, with the skin sterilized as per the ISSM guidelines for penile prosthesis implantation, thereby allowing primary repair of urethral injuries should they occur, and implantation in the same setting, without a higher risk of infection.

The study will involve 100 male patients undergoing aseptic surgery (regardless the procedure). Patients will be divided into two groups:

Group 1: control group, n=50 Group 2: Chlorhexidine group (Ch group), n=50 Pre-operatively, urethral instillation with Chlorhexidine gel will be performed for the Ch group, while for the control group, instillation will not be performed.

After conclusion of surgery and with the patient on the operative table, the following swabs will be obtained:

* A penile skin swab.
* A urethral swab. Skin and urethral swabs will be compared for bacterial colonization by culture and sensitivity, across the two groups.

DETAILED DESCRIPTION:
study design Comparative experimental (interventional) study Sample size

The study will involve 100 male patients undergoing aseptic surgery (regardless the procedure). Patients will be divided into two groups:

Group 1: control group, n=50 Group 2: Chlorhexidine group (Ch group), n=50

Pre-operatively, urethral instillation with Chlorhexidine gel will be performed for the Ch group, while for the control group, instillation will not be performed.

Chlorhexidine gel will be prepared according to an international product; Instillagel®, used prior to urethral catheterization as analgesic / anti-septic, with the following composition:

6ml of Instillagel® gel contain: 117.6mg lidocaine hydrochloride, 3.1mg chlorhexidine digluconate, 3.8mg methyl hydroxybenzoate (E218), 1.6mg propyl hydroxybenzoate (E216) 11ml of Instillagel® gel contain: 215.7mg lidocaine hydrochloride, 5.8mg chlorhexidine digluconate, 6.9mg methyl hydroxybenzoate (E218), 2.9mg propyl hydroxybenzoate (E216)

The other ingredients are:

Hyetellose, propylene glycol* (E 1520), sodium hydroxide and purified water. Intra-operatively, the Ch group will receive Chlorhexidine instillation again before surgery, while the control group will not.

For both groups, skin sterilization will be performed according to the ISSM "International Society of Sexual Medicine" guidelines for skin preparation before penile prosthesis surgery (Darren J. Katz et.al 2012)

After conclusion of surgery and with the patient on the operative table, the following swabs will be obtained:

* A penile skin swab.
* A urethral swab.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 20-50 years-old or older undergoing a sterile surgical procedure

Exclusion Criteria:

* Unwilling patient for this procedure
* Patients with history of urethral surgery, urinary calculi, urethral structure, or ongoing pyospermia, prostatitis or pyuria will be excluded, and so will be patients undergoing non-sterile surgeries such as abscess drainage.

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Bacterial colonization by culture and sensitivity | 4 days
  After conclusion of surgery and with the patient on the operative table, the following swabs will be obtained:
  * A penile skin swab.
  * A urethral swab. Skin and urethral swabs will be compared for bacterial colonization by culture and sensitivity, across the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Andrology department - Kasr El Aini Hospitals - Faculty of Medicine - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided